CLINICAL TRIAL: NCT06109675
Title: Nutritional Status Assessment of Pediatric Cystic Fibrosis Patients and Effect of Nutrition Education on Nutritional Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Merve Pehlivan, Phd(c), Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CyfNutEdu
Record Dates: First submitted 2023-10-19; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis in Children
Keywords: cystic fibrosis; nutrition education; nutritional status
MeSH Terms: conditions — Cystic Fibrosis | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental)
  Interventions: Behavioral: Nutrition Education
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Nutrition Education — All mothers in this group will be given 3 nutrition education sessions including detailed informations on Nutrition Therapy in Cystic Fibrosis. In addition to the education sessions, an informational booklet and a high-energy sample recipe booklet will be given.
  Arms: Education group

SUMMARY:
The goal of this clinical trial is to to assess the nutritional status of children diagnosed with cystic fibrosis between the ages of 2-14, to determine the changes in the nutrition education given to the mothers of the patients on the nutritional status of the children and the nutritional knowledge of the mothers, and to compare them with the control group.. The main questions it aims to answer are:

1. Will be better the nutritional status of children of mothers in the education group will be better compared to the control group?
2. Will the macro and micronutrient Recommended Dietary Allowance (RDA) and diet quality of children with cystic fibrosis in education group increase after nutrition education?
3. Will the nutrition knowledge test scores of mothers of children with cystic fibrosis in education group on "Nutrition in Cystic Fibrosis" increase after nutrition education?

Mothers of children diagnosed with cystic fibrosis will participate in the study as a result of the call of the Cystic Fibrosis Association in Turkey. Mothers participating in the study will be divided into 2 groups. While the mothers in the first group will be given nutrition education 3 times a week, 1 hour a day, no education session will be given to the mothers in the control group. The nutritional status and nutrient consumption of children in the training group and the control group will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Mothers included in the research must have responded to the KIFDER (Cystic Fibrosis Association in Turkey) call.
* Children of mothers included in the research must have been officially diagnosed with cystic fibrosis.
* Mothers included in the research mustn't receive any nutrition education beforehand.
* Children of mothers included in the research mustn't be regularly followed by a dietitian.

Exclusion Criteria:

* Children of mothers included in the research mustn't have a feeding tube.
* Children of mothers included in the research mustn't be diagnosed with any other disease known to affect growth.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Malnutrition rate in children with cystic fibrosis | Beginning of the study, 1st and 3rd months of the study
  According to the World Health Organisations (WHO) standarts; children who are more than 2 SD below the reference median are considered to be malnourished to be stunted, wasted or to be underweight. Children with measurements below 3 SD (a Z-Score of less than-3) are considered to be severely malnourished.
Malnutrition rate in children with cystic fibrosis | Beginning of the study, 1st and 3rd months of the study
  All children will also be evaluated according to the percentile recommendations in the guide of the European Cystic Fibrosis Society (ECFS). According to the ECFS guideline, those with height for age and BMI for age below the 50th percentile are classified as undernourished.

SECONDARY OUTCOMES:
The rate at which macronutrient and micronutrient consumption of children participating in the study meets the Recommended Dietary Allowance (RDA). | Beginning of the study, 1st and 3rd months of the study
  Recommended Dietary Allowance (RDA): Average daily level of intake sufficient to meet the nutrient requirements of nearly all (97-98%) healthy individuals; often used to plan nutritionally adequate diets for individuals.The macro and micronutrient RDA is determined by the Food and Nutrition Board of the National Academies of Sciences Engineering, and Medicine.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol Unıversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT06109675/Prot_000.pdf